CLINICAL TRIAL: NCT07033221
Title: Evaluation of the Effect of Bariatric Surgery on the Vestibular System in Obese Patients.
Brief Title: Vestibular Function in Obesity
Status: Recruiting | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Yusuf Emre ALTUNDAL, Assistant Professor, Istanbul Aydın University
Other Study IDs: 60/2025
Record Dates: First submitted 2025-05-24; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Vestibular Function Disorder; Balance Assessment; Balance Impairment; Sleeve Gastrectomy
Keywords: sleeve gastrectomy; balance in obese patients; vestibular function after sleeve gastrectomy; vestibulopathy in and obesity
MeSH Terms: conditions — Obesity; Vestibular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have demonstrated that obesity negatively affects the human vestibular system. However, whether improvement in vestibular function occurs following the resolution of obesity remains an area requiring further investigation. Therefore, the investigators aimed to assess and analyze vestibular system functions in patients scheduled for bariatric surgery, both before the surgery, after the surgery, and following significant weight loss.

Participants aged between 18 and 60 years who meet the inclusion criteria will be enrolled in the study. Initially, participants will undergo medical history assessment and Body Mass Index (BMI) measurement. The enrolled participants will be evaluated using the following tests at three different time points-preoperatively, at the 1st month postoperatively, and at the 6th month postoperatively: Video Head Impulse Test (vHIT), static posturography test, Berg Balance Scale, SF-12 Quality of Life Scale, and the Activity-specific Balance Confidence (ABC) Scale.

Although obesity has been shown to be associated with impaired postural balance, studies evaluating the direct effect of BMI on postural sway are limited. The aim of our study is to assess the vestibular system in obese patients before and after bariatric surgery. Through this, the investigators hope to contribute to the literature by providing balance assessments in individuals with obesity

ELIGIBILITY:
Inclusion Criteria:

1. The native language must be Turkish
2. The participant must be between the ages of 18-60
3. The participant must be suitable for bariatric surgery (BMI ≥40 kg/m2)
4. Not have any previous vestibular diagnosis
5. Not have any problems such as joints, muscles, or walking

Exclusion Criteria:

Individuals with additional disabilities, neurological problems, vestibulopathy, joint, muscle or walking disorders will not be included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants to be included in the study will be reached from patients who have applied to our hospital due to morbid obesity and are planned to undergo bariatric surgery in our hospital. Participants who meet the inclusion criteria and sign the Informed Voluntary Consent Form will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vestibular Function as Measured by Video Head Impulse Test (vHIT) | 12 months
  The vHIT assesses semicircular canal function by recording eye movements in response to brief, passive head rotations.
Change in Balance Performance Using Static Posturography | 12 months
  Objective measurement of postural sway and stability using a force platform system under various sensory conditions.

SECONDARY OUTCOMES:
Change in Functional Balance Measured by Berg Balance Scale (BBS) | 12 months
  The BBS is a 14-item scale evaluating balance during functional activities. Scores range from 0 to 56.
Change in Quality of Life as Measured by the SF-12 Health Survey | 12 months
  The SF-12 is a self-reported questionnaire assessing physical and mental health-related quality of life.
Change in Balance Confidence Measured by the Activity-specific Balance Confidence (ABC) Scale | 12 months
  Self-reported confidence in performing various daily activities without losing balance. Scores range from 0% to 100%.

OTHER OUTCOMES:
Obesity Status: Height, Weight, and Body Mass Index (BMI) | 12 months
  Anthropometric measurements taken using standard protocols. BMI calculated as weight (kg) divided by height (m²).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University Faculty of Medicine, Istanbul, Küçükçekmece, Turkey (Türkiye)